CLINICAL TRIAL: NCT03873285
Title: Development of a Genetic Analysis Method by Mendeliomes and Genomes in the Diagnosis of Genodermatoses and Rare Genetic Diseases With Cutaneous Expression
Brief Title: Method of Genetic Analysis in Genodermatoses
Acronym: GENODERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Center of Human Genetics - ULB in Brussels (Unknown); Interuniversity Institute of Bioinformatics in Brussels (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2018/Dermato/Genodermatose
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Genodermatosis; Rare Genetic Disease With Cutaneous Expression
Keywords: Genodermatosis; genetic; children
MeSH Terms: conditions — Skin Diseases, Genetic | interventions — Genome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genodermatosis patients (Experimental): Children between 0 to 18 years old with the presence of dermatological symptoms suggesting genodermatosis or presence of systemic symptoms in an undiagnosed patient associated with dermatological manifestations suggestive of a more rare genetic disorder with cutaneous expression
  Interventions: Genetic: Genetic diagnostic by mendeliome or genome

INTERVENTIONS:
Genetic: Genetic diagnostic by mendeliome or genome — For cases not explained by a mendeliomes: genome and transcriptome on fibroblast culture

SUMMARY:
The goal of the study is to develop a method of genetic diagnosis in two stages, by mendelioma then by genome and transcriptome on fibroblast culture, in genodermatoses and rare diseases with cutaneous expression in the child.

DETAILED DESCRIPTION:
Interventional multicenter prospective study. Patients will be examined by a dermatologist to describe and identify the various skin lesions Collaboration with the geneticist team: clinical examination for relevant cases Patient records will be consulted. Relevant medical information, biological examinations and other complementary examinations will be studied.

A blood sample (10 ml in EDTA tube) will be collected from the patient and his/her parents to store DNA for mediome and genome.

A written parental and child consent (if age-appropriate) will be obtained and a study information sheet will be signed. They will also sign the usual genetic consent request for mendeliome, genome and transcriptome on culture of fibroblasts.

A 4 mm punch skin biopsy (healthy or damaged depending on phenotype and indication) will be performed according to the standard technique.

The fibroblast culture will be performed routinely by the Genetics Center Transcriptome will be done according to the processes set up at the Genetics Center Mendeliome analysis

* Allow the analysis of 4000 rare disease genes
* Will be performed according to routine analyzes of the genetics lab
* Uses the Highlander tools (web)
* Use of de novo filters, autosomal recessive, heterozygous compound, X linked, strong variant (LOF and canonical splice sites)
* Use of rarer filters: exomic or gene deletion, splicing (+/- 12 base pairs around exons)
* In unexplained severe cases, a genome supplemented with the 10Xgenomics method and a transcriptome of fibroblasts will be realized. This double strategy afford to get a genome of high interpretative quality. Genome analysis by the 10Xgenomics method (https://www.10xgenomics.com )
* This method allows us to deconvolate haplotypes and allows the analysis of 16,000 other complementary genes and to obtain precisely defined structural variants.
* The transcriptome will better assess the genomic effects on gene expression.
* The genome and transcriptome will also assess the presence of deep intron mutations and their effect on splicing, and will be a sustainable resource for other long-term projects (analysis of non-coding regions, microRNAs, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Children between 0 to 18 years old
* Presence of dermatological symptoms suggesting genodermatosis
* Presence of systemic symptoms in an undiagnosed patient associated with dermatological manifestations suggestive of a more rare genetic disorder with cutaneous expression

Exclusion Criteria:

* Mosaicism
* Neurofibromatosis, all type
* Tuberous sclerosis
* Ichthyosis vulgaris
* Suspicion of somatic impairment (giant nevus)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Genetic diagnostic by mendeliome | At time of clinical diagnosis of genodermatosis
  Proportion of patients for whom a genetic diagnosis has been established using the mendeliome method. American College of Medical Genetics and Genomics. Diagnostic variants are classified as "pathogenic" or "probably pathogenic" variants.

SECONDARY OUTCOMES:
Genetic diagnostic by genome | At time of clinical diagnosis of genodermatosis
  Proportion of patients for whom a genetic diagnosis has been established using the genome method. American College of Medical Genetics and Genomics. Diagnostic variants are classified as "pathogenic" or "probably pathogenic" variants.
Genetic diagnostic by fibroblast transcriptome | At time of clinical diagnosis of genodermatosis
  Proportion of patients for whom a genetic diagnosis has been established using the fibroblast transcriptome method. American College of Medical Genetics and Genomics. Diagnostic variants are classified as "pathogenic" or "probably pathogenic" variants.
Relevance of dermatological symptoms | At time of clinical diagnosis of genodermatosis
  Correlation between dermatological signs and symptoms and a genetic diagnosis established by the mendelioma, genome and transcriptome method

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Salik, MD, Principal Investigator — Hôpital Universitaire Des Enfants Rein Fabiola
Locations (1):
- Hôpital Universitaire Des Enfants Rein Fabiola, Brussels, Belgium